CLINICAL TRIAL: NCT06896539
Title: Tele-health for Contraceptive Counselling - a Randomized Controlled Trial of Contraceptive Counselling Via Tele-health Compared to Standard Routine on the Effects of Choice and Uptake of LARC
Brief Title: Telemedicine for Contraceptive Counselling- An Open Randomized Controlled Trial
Acronym: Tele-prev
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Örebro University, Sweden (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-08130-02
Record Dates: First submitted 2025-03-12; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Unintended Pregnancy Prevention
Keywords: Telemedicine; Contraception; Unintended pregnancy; Counselling
MeSH Terms: interventions — Telemedicine; Counseling

STUDY DESIGN:
Intervention Model Description: Open randomized non-inferiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counselling through Telemedicine (Experimental): Contraceptive counselling using LOWE methodology via telemedicine (video calls).
  Interventions: Other: Telemedicine
- Contraceptive counselling via in-person visit (Other): Contraceptive counselling using the LOWE methodology via in-person visit.
  Interventions: Other: Counselling in person visit

INTERVENTIONS:
Other: Telemedicine — Contraceptive Counselling using the "LOWE Method" and through Tele Health, Video Call with Midwife.
  Other Names: Tele health
  Arms: Counselling through Telemedicine
Other: Counselling in person visit — Contraceptive Counselling using the "LOWE Method". In-person visit with midwife at Maternal Health Clinic.
  Other Names: In person
  Arms: Contraceptive counselling via in-person visit

SUMMARY:
Protocol Summary:

Sweden has high unintended pregnancy rates, increasing unmet contraceptive needs, and the highest repeat abortion rate in the European Union. Effective contraceptive counseling can improve satisfaction, empower correct use, and increase uptake of long-acting reversible contraceptives (LARC), potentially reducing unintended pregnancies.

Research has explored ways to enhance contraceptive counseling, focusing on increasing LARC use. Interventions that improve access, remove financial barriers, and enhance method-specific knowledge-especially regarding effectiveness-have led to higher LARC adoption and fewer unintended pregnancies and abortions.

The COVID-19 pandemic significantly increased tele-health use for contraceptive counseling. Studies suggest tele-health expands appointment availability, reduces geographic barriers, and improves access to reproductive care, particularly in low-resource populations. However, few studies have examined tele-health's impact on contraceptive counseling, uptake, and satisfaction compared to in-person visits, particularly in Sweden. Before tele-health can be established as a viable family planning option, its counseling quality and impact on LARC adoption must be assessed.

Study Aims:

To determine whether the choice of LARC after tele-health (video) counseling is comparable to in-person counseling with a midwife, using structured contraceptive counseling in both groups.

To assess whether LARC uptake three months post-counseling is similar between women who received tele-health vs. in-person counseling.

This study will provide valuable insights into tele-health's role in contraceptive counseling and its potential to improve access to family planning services.

DETAILED DESCRIPTION:
Unintended pregnancies and unmet contraceptive needs remain critical global reproductive health concerns. Sweden has a high unintended pregnancy rate and the highest repeat abortion rate in the Eropean Union (EU). In 2021, approximately 33,700 abortions were reported in Sweden, equating to 18 per 1,000 women aged 15-44 . Beyond personal challenges, unintended pregnancies impose significant healthcare costs, estimated at 448 million Swedish Crones annually.

With the mean age for first-time mothers exceeding 30 years in most European countries, many women require effective contraception for extended periods. Contraceptive effectiveness is measured using the Pearl Index (PI), which reflects pregnancy rates per 100 women per year under "perfect use" versus "typical use." Long-acting reversible contraception (LARC), including intrauterine devices (IUDs) and contraceptive implants, minimizes user-dependent failure, making it the most effective and satisfactory method . A 5% increase in LARC use among Swedish women could prevent 3,500 unintended pregnancies annually, saving over SEK 70 million.

Increasing contraceptive prevalence and LARC adoption can reduce unintended pregnancies. Sweden's 2014 national contraception guidelines emphasized protecting fertility and preventing unintended pregnancy. In 2020, the Swedish Family Planning Reference Group set goals for LARC adoption: 40% after primary care visits and 60% post-abortion. A 2017 survey showed 71% of Swedish women used contraception, with LARC at 30.9%, an increase from 2013. However, unmet contraceptive needs rose from 9% in 2013 to 15% in 2017. Women using oral contraceptives, patches, or vaginal rings had a 20-fold higher failure rate than LARC users. A 2022 internet survey reported lower LARC use (19.8%) but confirmed high unmet contraceptive needs. A 5,000-woman cohort study found 84% satisfaction with LARC after one year, versus 53% for non-LARC methods.

Structured Contraceptive Counselling No universally effective contraceptive counseling model exists, and provider bias can affect recommendations. Swedish surveys highlight contraceptive effectiveness as a top priority for patients, yet oral contraceptives remain the most used method in Europe and the U.S.

Efforts to improve contraceptive counseling, particularly for LARC promotion, have shown that removing financial barriers and increasing method-specific knowledge improves LARC uptake and reduces unintended pregnancies. A cluster-randomized trial in Stockholm with 1,364 participants at youth clinics, abortion clinics, and maternal health centers evaluated the structured contraceptive counseling method "The LARC Forward Counselling method (LOWE)". This approach included a 7-minute educational video, four key questions, a tiered effectiveness chart, and a demonstration box with contraceptive models. Women receiving this structured counseling were more likely to choose LARC (40.6% vs. 30.3% in standard counseling). The method was equally effective among migrants, reduced repeat unintended pregnancies among abortion patients, and was rated time-neutral and beneficial by healthcare providers.

Tele-Health and Contraceptive Counselling The World Health Organization (WHO) defines tele-health as "the delivery of health care services, where patients and providers are separated by distance". Tele-health can include phone consultations, video calls, mobile applications, and email.

Studies suggest tele-health expands healthcare capacity, increases appointment availability, and reduces geographic and socioeconomic barriers to reproductive care. A study of 18,000 women found that pre-abortion contraceptive counseling via tele-health led to higher LARC uptake compared to in-person counseling during abortion consultations.

Text message-based interventions have also been explored to improve contraceptive adherence and continuation. One study showed that daily educational text messages significantly increased six-month oral contraceptive continuation rates. Two randomized controlled trials demonstrated the effectiveness of text reminders in improving adherence to oral contraceptives and injectable depo contraceptives.

This research highlights tele-health's potential to improve contraceptive counseling access, reduce unintended pregnancies, and enhance LARC adoption.

In conclusion, more research is needed to study if tele-health can be used in general settings and not only in selected groups. There is also a need to further understand patient´s experience of tele-health for contraceptive counselling to determine whether it can meet patients' needs and if contraceptive counselling through tele-health, effects the uptake of LARC in a Swedish context.

Study design: An open randomized, controlled, non-inferiority trial.

Study objects: Women contacting maternal health clinics (MHC) for contraceptive counselling.

Sample size: 772 participants.

Data will be collected from April 2025 June. 2027. Inclusion time- 2 years.

Method:

Randomized controlled non-inferiority trial (RCT). All data collection will be performed using the electronic data collection program Smart Trial.

Eligible women who contact a midwife at a maternal health clinic (MHC) for contraceptive counselling (CC) will be informed about the study verbally and invited to participate. The written study information will include contact information to the responsible researchers to answer any questions, as well as a link to the informed consent form. Women who consent to participate will get an appointment, not specifying if the appointment will be digital or in person during a regular visit. After written consent, the Smart Trial randomization plug-in will automatically allocate participants in a 1:1 ratio to receive structured contraceptive counselling either via telehealth video (intervention) or via in-person visit (control).

Before the counselling session, the participant will receive a first survey of background variables including socio-demographic variables such as BMI, educational level, country of birth, and contraceptive and reproductive history. Women who are randomized to tele-health (video counselling) and choose combined pill/ patch will be asked to register blood pressure after the appointment. Participants with blood pressure over 140/90 will be asked to contact a health care clinic according to standard guidelines.

After completing the first survey, the participants will be linked to the educational video which is to be seen prior to the rest of the counselling (see description of structured contraceptive counselling above). visit.

The tele-health counselling will be provided using a virtual care platform. All patient data is handled following General Data Protection Regulation and the Patient Data Act.

At the end of the counselling, the midwife will complete a survey to register the contraceptive choice. Participants in both the intervention and control group, choosing LARC will receive a second, in person appointment for placement of the method.

After the counselling, participants will receive a second survey with questions regarding the experience with the contraceptive counselling, questions about participant autonomy, and also questions about the LOWE methodology.

Follow-up surveys will be sent to participants at 3 and 12, months after the counselling, to collect data on method initiation continued use satisfaction, method switching, pregnancies and outcomes of pregnancies. Medical records will be scrutinized for pregnancies and pregnancy outcomes within 24 months. Data will be collected anonymised.

Analyse:

Data will be analyzed using descriptive statistics. T-test and Mann-Whitney u-test will be used where appropriate. Logistic regression models will be used to assess association between demographic characteristics and LARC choice and to assess factors related to use of contraception and risk of subsequent pregnancy and abortions.

Statistical power RCT with non-inferiority design. The number of users of LARC vary widely between studies. Two recent Swedish publications have reported substantially different figures; 19.8% vs 30.7% and consequently it is difficult to adequately estimate the number of women who will chose LARC. Several other studies have reported similar figures.

The hypothesise is that 25% of all women will chose LARC and that the number is not lower in the intervention group. Given a non-inferiority limit of 10% (Δ), 90% power (1-β) and 5% significance level (α) the study population need to consist of 644 women, 322 in each group. To compensate for an estimated 20% loss to follow-up the investigators aim to include 772 participants.

Ethical considerations:

In the present study, the data will be handled and analysed anonomysed and the results will not be presented on an individual level. The code key will be stored locked and only available for the responsible researcher. Written consent for the use of medical records will be obtained in accordance with the Personal Data Act.

The study will be performed according to the Declaration of Helsinki. Patients will receive oral and written information emphasising that participation is voluntary, before giving their consent to participate.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 16-40 years
* Primary reason for use of contraception being pregnancy prevention
* Not having pregnancy intentions within 6 months.
* Sufficient language skills to understand the study information available in Swedish and English.

Exclusion Criteria:

* Women in need for contraceptive method for medical reasons other than protection against unintended pregnancy.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 772 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in LARC use | From enrollment to 12 months.
  Difference in proportion of women choosing LARC among participants receiving structured contraceptive counselling via telehealth (intervention) compared to in-person visit (control).

CONTACTS AND LOCATIONS:
Overall Officials: Jan Brynhildsen, PhD, Principal Investigator — Örebro Universitet, Region Örebro

IPD SHARING:
Plan to Share IPD: No
According to Swedish law.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT06896539/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT06896539/ICF_001.pdf